CLINICAL TRIAL: NCT03107858
Title: The Effect of Norepinephrine Versus Dopamine in Renal Transplant Recipients on Postoperative Graft Function
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Abdel Kader Ahmed Mohammed Elkadi, Specialist, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NorepivsDopamine
Record Dates: First submitted 2017-03-24; First posted 2017-04-11 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Renal Transplant
MeSH Terms: interventions — Norepinephrine; Dopamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Norepinephrine (Active Comparator)
  Interventions: Drug: Norepinephrine
- Dopamine (Active Comparator)
  Interventions: Drug: Dopamine

INTERVENTIONS:
Drug: Norepinephrine — Norepinephrine infusion will be used at a starting dose of 0.05μg/kg/min. Dose range: 0.05 -0.15 μg/kg/min. Infusion will be started with arterial decamping and continues till 24 hours postoperative
  Arms: Norepinephrine
Drug: Dopamine — Dopamine infusion will be used at a starting dose of 5μg/kg/min. Dose range: 5 -15 μg/kg/min. Infusion will be started with arterial decamping and continues till 24 hours postoperative
  Arms: Dopamine

SUMMARY:
Renal transplantation is now recognized as a treatment of choice for patients with chronic renal failure with end-stage renal disease. Renal transplantations are associated with better quality of life, better cost/benefit ratio, and possibly longer survival. Significant changes in blood pressure are common throughout the surgical procedure for kidney transplantation. All efforts are made to maintain an appropriate level of blood pressure by using an adequate intravascular volume and vasopressor administration. All efforts are made to maintain an appropriate level of blood pressure by using an adequate intravascular volume and vasopressor administration. All efforts are made to maintain an appropriate level of blood pressure by using an adequate intravascular volume and vasopressor administration. All efforts are made to maintain an appropriate level of blood pressure by using an adequate intravascular volume and vasopressor administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for a living donor kidney transplantation

Exclusion Criteria:

* Patients (less than 18 years old)
* Patients' refusal of consenting for enrolment in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
serum creatinine | four hours postoperatively
  postoperative

SECONDARY OUTCOMES:
blood urea | four hours postoperatively
  postoperative
urine output | over 24 hours
  postoperative
renal artery diameter | four hours postoperatively
  Measured postoperative through renal artery Doppler
renal artery blood flow | four hours postoperatively
  Measured postoperative through renal artery Doppler

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided